CLINICAL TRIAL: NCT01663181
Title: Pain-perception During Outpatient cystoscopy-a Prospective Controlled Study
Status: Completed | Type: Observational
Sponsor: Medical University of Vienna (Other)
Responsible Party: Principal Investigator, Wolfgang Umek, MD, ao.Univ.Prof.Dr.univ.med, Medical University of Vienna
Other Study IDs: 413/2009
Record Dates: First submitted 2012-08-05; First posted 2012-08-13 (Estimated); Last update posted 2022-04-12 (Actual); Status verified 2022-04

CONDITIONS: Urinary Incontinence; Overactive Bladder; Pelvic Organ Prolapse; Recurrent Urinary Tract Infections
MeSH Terms: conditions — Urinary Incontinence; Urinary Bladder, Overactive; Pelvic Organ Prolapse; Urinary Tract Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- urogynecologic patients undergoing outpatient cystoscopy
- urogynecologic patients undergoing outpatient-urodynamics

SUMMARY:
At an academic tertiary referral center, patients with pelvic floor dysfunction, scheduled for outpatient cystoscopy or urodynamic testing will be asked to participate in the study. Patients will be called one day after the examination and will be asked about pain and their general state of health.

The purpose of this study it to investigate pain perception in urogynecologic patients during outpatient cystoscopy and compare it with pain perception during outpatient urodynamic. The investigators will also investigate the difference between anticipated and actual pain perception. The investigators will test the null hypothesis that there is no difference in patients´ pain perception between outpatient cystoscopy and urodynamic testing. The secondary hypothesis will be that there is no difference between patients´ anticipated amount of pain and the actually experienced pain during cystoscopy and urodynamic testing.

According to power calculation, a sample size of 52 patients per group will be needed to detect a 2 cm difference in pain scores on the VAS - judged as a clinically significant difference - with 95% power and a two-sided significance level of 0.05.

Exclusion criteria are: age ≤ 18 years, insufficient ability to understand German, pregnancy and the participation in another clinical study at the same time.

ELIGIBILITY:
Inclusion Criteria:

* women undergoing cystoscopy or urodynamic testing at an academic tertiary referral center.

Exclusion Criteria:

* age ≤ 18 years
* insufficient ability to understand German
* pregnancy
* participation in another clinical study at the same time

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: women, aged >= 18 years with pelvic floor dysfunction, undergoing diagnostic work-up at a tertiary referral center for urogynecologic conditions
Sampling Method: Non-Probability Sample
Enrollment: 109 (Actual)
Dates: Start 2009-05; Primary Completion 2010-02 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
subjective pain perception immediately after examination as measured by a standard visual analog scale | immediately after examination (zero to ten minutes after completing cystoscopy or urodynamics)
  patients are assessed at three points in time:
  1. zero to ten minutes before undergoing examination
  2. zero to ten minutes after undergoing examination
  3. 24 hours after undergoing examination

SECONDARY OUTCOMES:
difference between anticipated pain and actual pain perception | immediately before and immediately after the examination (zero to ten minutes after undergoing examination)

CONTACTS AND LOCATIONS:
Overall Officials: Wolfgang Umek, Prof, Principal Investigator — Medical University Vienna Austria
Locations (1):
- Medical University Vienna, Vienna, Austria